CLINICAL TRIAL: NCT07133841
Title: Validity of Thermal Imaging in Injury Risk Assessment in Volleyball Players: A Comparative Analysis With Performance Tests
Brief Title: Validity of Thermal Imaging in Injury Risk Assessment in Volleyball Players
Status: Recruiting | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Begum Kara Kaya, Assistant Professor, Biruni University
Other Study IDs: BAP
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-08

CONDITIONS: Athletes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pre-Season Assessments — Pre-Season Assessments including performance based tests and thermal imaging.

SUMMARY:
Although studies in the literature have used thermography for injury prevention and performance monitoring in various sports, no systematic validation of the method has been conducted in volleyball players. This study aims to determine whether thermography is a reliable and standardized tool for injury risk assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 18 and 30 years old
* Volunteer to participate in the study
* For women, be in the follicular phase of their menstrual cycle
* Be able to understand and speak Turkish
* Be in the team's preseason
* Have been playing volleyball on the team at the amateur/professional level for at least one year
* Have no ongoing musculoskeletal problems that prevent exercise

Exclusion Criteria:

* Continuing active rehabilitation
* Body mass index ≥ 30 kg/m2
* Having an active infectious/inflammatory disease (rheumatoid arthritis, sacroiliitis, bursitis, synovitis, etc.)
* Having consumed/taken coffee, alcohol, cigarettes, analgesics, anti-inflammatory medications, etc., within the 24 hours prior to the evaluation.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: İstanbul/Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Thermal Camera Imaging | 2 weeks
Vertical Jump Test | 2 weeks
Dynamic Balance Assessment | 2 weeks

SECONDARY OUTCOMES:
Functional Movement Screening | One week
Muscle Strength Assessment | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No